CLINICAL TRIAL: NCT00831961
Title: Prospective, Randomized, Observational Cohort Study of Antibiotic Resistance After Repeated Application of Topical Antibiotics
Brief Title: Antibiotic Resistant Patterns of Conjunctival and Nasophayngeal Flora After Repeated Exposure to Topical Antibiotics
Acronym: ARCaNE
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Stephen J. Kim, MD, Associate Professor of Ophthalmology, Vanderbilt University
Other Study IDs: 090020
Record Dates: First submitted 2009-01-28; First posted 2009-01-29 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Age-related Macular Degeneration
Keywords: Antibiotic resistance, Conjunctival flora, Intravitreal injections
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: Patients randomized to gatifloxacin (Zymar)
  Interventions: Procedure: Conjunctival and nasopharyngeal bacteria cultures
- 2: Patients randomized to moxifloxacin (Vigamox)
  Interventions: Procedure: Conjunctival and nasopharyngeal bacteria cultures
- 3: Patients randomized to ofloxacin (Ocuflox)
  Interventions: Procedure: Conjunctival and nasopharyngeal bacteria cultures
- 4: Patients randomized to azithromycin (AzaSite)
  Interventions: Procedure: Conjunctival and nasopharyngeal bacteria cultures

INTERVENTIONS:
Procedure: Conjunctival and nasopharyngeal bacteria cultures — Conjunctival and nasopharyngeal bacteria cultures

SUMMARY:
Repeated exposure to topical antibiotics may alter the normal bacteria on the eye and in the nose and increase rates of resistance. This study will determine whether repeated short-term exposure to topical antibiotic drops which are commonly prescribed after eye injections to reduce the chance of infection increase rates of resistant bacteria which are normally found on the eye and in the nose.

We hypothesis that certain commercially available antibiotics may increase rates of bacteria resistance more so than others.

DETAILED DESCRIPTION:
Introduction

The treatment of neovascular age-related macular degeneration (AMD) with anti-vascular endothelial growth therapy (ranibizumab and bevacizumab, Genentech, South San Francisco, CA) requires repetitive and often long-term intraocular injections and has raised concern about increasing rates of endophthalmitis. Endophthalmitis remains one of the most feared complications in ophthalmology and despite early detection and intervention can result in substantial morbidity. Recent multicenter clinical trials of anti-vascular endothelial growth therapy have reported endophthalmitis rates of 1.0% to 1.9% per patient treated (during a 6 month to 2 year period of follow-up). Consequently, topical antibiotics are routinely prescribed after intraocular injections, although no published study to date has proven their efficacy in preventing post-injection endophthalmitis. 1,2

Of increasing concern, however, are reports of growing resistance of normal ocular flora to commonly employed antibiotic classes including macrolides, aminoglycosides, and 3rd generation fluoroquinolones.3-5 The recent availability of 4th generation fluoroquinolones: gatifloxacin 0.3% (Zymar, Allergan Pharmaceuticals, Irvine, Calif) and moxifloxacin 0.5% (Vigamox, Alcon Fort Worth, TX) has notably enhanced our armamentarium and are widely used due to their greater potency. Not surprisingly however, recent reports have begun to surface documenting emerging resistance to these 4th generation fluoroquinolones as well.6,7

The practice of short-term and repeated exposure of ocular flora to antibiotics, as is the case after intraocular injections for AMD, may facilitate antibiotic resistance. However, no study to date has evaluated resistance patterns of ocular or nasopharyngeal flora in response to repeated applications of topical antibiotics over time.

Therefore, this study will attempt to monitor long-term resistance patterns of conjunctival and nasopharyngeal flora in patients with AMD who are repeatedly exposed to different commercially available antibiotics after intraocular injections.

Objective of the Research Study:

To determine changes in ocular and nasopharyngeal flora after repeated exposure to topical antibiotics.

Research Hypothesis:

Rpeated use of topical antibiotics may alter normal ocular and nasopharyngeal flora and may increase resistance to commonly employed antibiotics.

Study Design: Prospective, randomized, observational cohort study

Specific Goals of the Study:

1. Establish baseline susceptibility and resistance patterns of normal conjunctival and nasopharyngeal flora of patients with choroidal neovascularization.
2. Monitor changes in normal conjunctival and nasopharyngeal flora after repeated exposure to topical antibiotics over a 2 year period.
3. Determine patterns of antibiotic resistance of conjunctival and nasopharyngeal flora after repeated exposure to topical antibiotics.

Previous Studies: none

Methods

The Vanderbilt University Institutional Review Board will approve this study and the study will comply with all aspects of the Health Insurance Portability and Accountability Act.

All adult patients with choroidal neovascularization (CNV) due to AMD or other causes in 1 eye and planned treatment with intraocular injections of either ranibizumab or bevacizumab, will be eligible. Patients will be excluded if they are younger than 18, are taking concurrent topical or systemic antibiotics, have active ocular infection, or have a history of use of topical antibiotics for any indication within the previous 3 months.

Patients identified with CNV after complete ophthalmic examination and who agree to participate will be asked to return ≥ 24 hours later for their planned injection in order to minimize contamination from topical anesthetic and mydriatic drops.

Patients will be assigned to 1 of 4 commercially available antibiotics at the initial study visit: ofloxacin 0.3% (Ocuflox, Akorn Inc., Somerset, NJ), azithromycin 1% (AzaSite, Inspire Pharmaceuticals, Inc. Durham, NC), gatifloxacin 0.3%, or moxifloxacin 0.5% and will use only their assigned antibiotic during and after all injections for the entire duration of the study.

Conjunctival cultures (from the lower fornix) of both eyes and nasopharyngeal cultures from the same side as the eye to be treated will be taken with sterile cotton tip applicators and calcium alginate swabs, respectively before the application of any topical medications. The cultures will be obtained in standardized fashion with every effort made to minimize contamination from the lids, lashes, or skin.

All intravitreal injections will be performed in accordance with the standard protocol of each individual treating retina specialist using sterile technique. Patients will start using their assigned antibiotic beginning on the day of their injection and continue for the next 4 consecutive days.

Conjunctival culture swabs will be transported to the microbiology laboratory using the BBLTM CultureSwabTM (Becton, Dickinson and Company, Sparks, MD 21152) transport system and then inoculated onto blood agar plates and incubated at 37°C for 3 days. All blood agar plates will be incubated in a microaerophilic environment. Blood agar cultures will be deemed positive if 1 or more colony forming units are observed. Nasopharyngeal swabs will be directly inoculated on blood agar plates and transported to the microbiology laboratory and processed as above.

To test resistance, the Kirby-Bauer disc diffusion technique will be conducted in accordance with the guidelines of National Committee for Clinical Laboratory Standards.

The following antibiotics will be tested for resistance on all positive cultures: penicillin, cefazolin, ceftazidime, imipenem, gentamicin, tobramycin, erythromycin, azithromycin, ciprofloxacin, ofloxacin, levofloxacin, gatifloxacin, moxifloxacin, doxycycline, and vancomycin.

All patients will return in 4 weeks and cultures will be retaken in the exact same fashion as above. If further injections are planned, the above protocol will be repeated until the end of the study.

Sample Size

Exact sample size calculations are difficult given the absence of reference data. We plan to follow patients for 2 years and anticipate requiring 10 patients for each antibiotic arm. We anticipate having 6 culture results per patient during the first year of follow-up and assume a 20% loss of follow-up. Thus, we plan to recruit a total of 48 participants.

Statistics

Descriptive statistics including mean and standard deviation will be calculated for case characteristics. Group comparisons will be performed with the Wilcoxon rank-sum test and chi-square test. A P value < 0.05 will be considered significant.

Study Withdrawal: patients will be reminded at every visit that they can discontinue the study at any time.

Patient information: all patient data will be recorded and retained using non-identifiers.

ELIGIBILITY:
Inclusion Criteria:

* age greater than 18 with choroidal neovascularization with planned treatment with intravitreal injections

Exclusion Criteria:

* Use of topical antibiotics for any reason within 3 months, current use of systemic or topical antibiotics, known allergies to gatifloxacin, moxifloxacin, ofloxacin, and azithromycin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients age greater than 18 with choroidal neovascularization with planned treatment with intravitreal injections.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2009-01; Primary Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Establish baseline susceptibility and resistance patterns of normal conjunctival and nasopharyngeal flora of patients with choroidal neovascularization. | 2 years
Monitor changes in normal conjunctival and nasopharyngeal flora after repeated exposure to topical antibiotics over a 2 year period. | 2

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Kim, MD, Principal Investigator — Vanderbilt University Department of Ophthalmology
Locations (1):
- Vanderbilt Eye Institute, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Kim SJ, Toma HS. Antimicrobial resistance and ophthalmic antibiotics: 1-year results of a longitudinal controlled study of patients undergoing intravitreal injections. Arch Ophthalmol. 2011 Sep;129(9):1180-8. doi: 10.1001/archophthalmol.2011.213. PMID 21911665